CLINICAL TRIAL: NCT04643392
Title: The Effects of Complex Decongestive Physiotherapy Applications on Upper Extremity Circumference and Volume in Patients With Lipedema
Brief Title: Physiotherapy Applications in Upper Extremity Lipedema
Status: Completed | Type: Observational
Sponsor: Yuksek Ihtisas University (Other)
Responsible Party: Principal Investigator, Melek Volkan Yazici, Principal Investigator, Yuksek Ihtisas University
Other Study IDs: YIU
Record Dates: First submitted 2020-11-18; First posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Lipedema
Keywords: Upper extremity lipedema; Lymphatic drainage
MeSH Terms: conditions — Lipedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Lipedema: Participants who were diagnosed with upper extremity lipedema by a lymphologist.
  Interventions: Procedure: Complex decongestive physiotherapy

INTERVENTIONS:
Procedure: Complex decongestive physiotherapy — Each patient received a treatment protocol of Complex decongestive physiotherapy for 5 days a week until they were discharged from the clinic. All patients fully completed all components of the treatment routine daily. The treatment was performed by a physiotherapist who was certified with Manual Lymph Drainage Combined Decongestive Physiotherapy. After the daily treatment protocol was completed, patients wore standard or individually sized compression grade II or III medical compression stockings for the rest of the day.

SUMMARY:
Lipedema which causes excessive accumulation of fat in the subcutaneous tissue, is a rare, progressive disease. This disease generally affects women, following puberty or early adulthood and usually results in the slow increase of the circumference of the legs and/or arms, bilaterally. In a typical presentation of lipedema, the enlargement of the lower extremities is disproportionately greater than that of the trunk and upper extremities When first described in 1940, lipedema was thought to exclusively affect the lower extremities. However, as the disease has been recognized over the years, lipedema has been reported to affect the upper extremities. Upper extremity lipedema, with no involvement of the lower extremities is an extremely rare incident.

DETAILED DESCRIPTION:
Due to the hypertrophy in adipose tissue, the link between lymphatic dysfunction and the progression to lipo-lymphedema, lipedema is conservatively treated with physiotherapy, manual lymph drainage and compression, also known as complex decongestive physiotherapy. Furthermore, the consensus of the International Society of Lymphology has stated that intermittent pneumatic compression is an optional treatment which may be applied as an adjuvant therapy to complex decongestive physiotherapy. All participants included in the study were included in a treatment protocol consisting of complex decongestive physiotherapy and intermittent pneumatic compression. The Perometer was used in the measurement of upper extremity volume and circumference before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* being between the ages of 18-65,
* having a diagnosis of upper extremity lipedema
* being willing to participate in the study

Exclusion Criteria:

* accompanying diagnosis of lymphedema,
* deep vein thrombosis
* disease which causes edema in the upper extremities

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between the age of 18-65 who have lipedema affecting the upper extremities and no accompanying diagnosis of lymphedema, deep vein thrombosis or any disease which causes edema in the upper extremities.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2020-05-04 (Actual)

PRIMARY OUTCOMES:
Limb Circumference | Change from baseline circumference at 4 weeks
  For every patient, the circumference measurements of the upper limbs were measured with the Perometer.
Limb Volume | Change from baseline volume at 4 weeks
  For every patient, the volume measurements of the upper limbs were measured with the Perometer.

CONTACTS AND LOCATIONS:
Overall Officials: Melek Volkan-Yazici, PT. PhD, Principal Investigator — Yuksek Ihtisas University; Murat Esmer, PT. MSc, Study Director — Gazi University
Locations (1):
- Yuksek Ihtisas University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Volkan-Yazici M, Esmer M. Reducing Circumference and Volume in Upper Extremity Lipedema: The Role of Complex Decongestive Physiotherapy. Lymphat Res Biol. 2022 Feb;20(1):71-75. doi: 10.1089/lrb.2020.0128. Epub 2021 Apr 5. PMID 33798399